CLINICAL TRIAL: NCT00718549
Title: A Randomized, Open Label Study to Assess the Effect of Maintenance Treatment With Mabthera (Rituximab) Versus No Treatment, After Induction Treatment With Rituximab, Cladribine and Cyclophosphamide (RCC) on Progression-Free Survival in Previously Untreated Patients With Progressive B-Cell Chronic Lymphocytic Leukemia
Brief Title: A Study to Assess the Effect of Maintenance Treatment With Rituximab Versus No Treatment in Participants With Progressive B-Cell Chronic Lymphocytic Leukemia (CLL)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML21283; 2008-001140-39
Record Dates: First submitted 2008-07-16; First posted 2008-07-18 (Estimated); Results first posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2017-11

CONDITIONS: Lymphocytic Leukemia, Chronic
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Cladribine; Cyclophosphamide; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Induction: Rituximab, Cladribine, Cyclophosphamide (Experimental): Participants will receive rituximab at a dose of 375 milligrams per meter squared (mg/m^2) as intravenous (IV) infusion on Day 1, cladribine at a dose of 0.12 milligrams per kilogram per day (mg/kg/day) as IV infusion on Days 2-4, and cyclophosphamide at a dose of 250 mg/m^2/day as IV infusion over 15-30 minutes on Days 2-4 in Cycle 1. Then, rituximab at a dose of 500 mg/m^2 as IV infusion on Day 1, cladribine at a dose of 0.12 mg/kg/day as IV infusion on Days 2-4, and cyclophosphamide at a dose of 250 mg/m^2/day as IV infusion over 15-30 minutes on Days 2-4 will be administered in Cycles 2-6. Each cycle will be of 28 days in duration.
  Interventions: Drug: Cladribine; Drug: Cyclophosphamide; Drug: Rituximab
- Maintenance Arm: Rituximab (Experimental): Participants with PR or CR after induction phase who will be randomized to maintenance arm will receive rituximab treatment for 8 cycles. Twelve weeks after the last induction cycle, participants will receive rituximab at a dose of 375 mg/m^2 as IV infusion on Day 1 of each 12-week cycle until disease progression (up to approximately 96 weeks).
  Interventions: Drug: Rituximab
- Observation Arm: No Intervention (No Intervention): Participants with PR or CR after induction phase who will be randomized to observation arm will not receive any intervention. Participants will be assessed every 4-weeks for the first 12 weeks and every 12-weeks afterwards up to 96 weeks.

INTERVENTIONS:
Drug: Cladribine — Cladribine will be adminiatered at a dose of 0.12 mg/kg/day as IV infusion on Days 2-4 of each 28-day cycle during induction phase.
  Arms: Induction: Rituximab, Cladribine, Cyclophosphamide
Drug: Cyclophosphamide — Cyclophosphamide will be administred at a dose of 250 mg/m^2/day as IV infusion over 15-30 minutes on Days 2-4 of each 28-day cycle during induction phase.
  Arms: Induction: Rituximab, Cladribine, Cyclophosphamide
Drug: Rituximab — Rituximab will be administered at a dose of 375 mg/m^2 as IV infusion on Day 1 of Cycle 1 and at a dose of 500 mg/m^2 as IV infusion on Day 1 of Cycles 2-6 during induction phase. Rituximab will be administered at a dose of 375 mg/m^2 as IV infusion on Day 1 of each 12-week cycle during maintenance phase.
  Other Names: MabThera
  Arms: Induction: Rituximab, Cladribine, Cyclophosphamide; Maintenance Arm: Rituximab

SUMMARY:
This study will assess the effect of maintenance treatment with rituximab in comparison with observation period (no treatment), in participants with progressive B-cell CLL who have had previous first-line induction treatment with rituximab, cladribine and cyclophosphamide (RCC regimen). After 6 months of RCC induction therapy, participants will be randomized either to receive maintenance treatment with rituximab or to receive no treatment (observation only) for 96 weeks. Participants completing maintenance/observation period will be followed-up for approximately 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Immunologically confirmed diagnosis of B-cell CLL
* Rai stage I-IV disease with evidence of progression
* No previous chemotherapy, radiotherapy, or immunotherapy for B-cell CLL
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2

Exclusion Criteria:

* Active secondary malignancy or transformation to aggressive lymphoma
* Medical condition requiring chronic use of oral corticosteroids at a dose of 1 mg/kg or 60 mg/m^2 over 2 weeks
* Prior treatment with interferon, rituximab or another monoclonal antibody, immunosuppressive treatment or radiotherapy before inclusion to the study
* History of other malignancies within 2 years before study entry, except for dequately treated carcinoma in situ of the cervix; basal or squamous cell skin cancer; low grade, early stage localized prostate cancer treated surgically with curative intent; good prognosis ductal carcinoma in situ (DCIS) of the breast treated with lumpectomy alone with curative intent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2009-07-21 (Actual); Primary Completion 2015-09-14 (Actual); Study Completion 2015-09-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- City Clinical Hospital #9, Minsk, Belarus
- Poland (5):
  - Medical University, Independent Public Clinical Hospital; Dept. of Hematology, SPSK, Bialystok
  - Szpital Uniwersytecki W Krakowie; Klinika Hematologii, Krakow
  - Medical University School; Dept. of Haematology, Lodz
  - Istytut Hematologii i Transfuzjologii; Hematologia, Warsaw
  - Medical Uni of Wroclaw; Hematology, Wroclaw

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 136 participants were screened, out of which 128 participants were enrolled in this study.
Groups:
- Induction: Rituximab, Cladribine, Cyclophosphamide: Participants received rituximab at a dose of 375 milligrams per meter squared (mg/m^2) as intravenous (IV) infusion on Day 1, cladribine at a dose of 0.12 milligrams per kilogram per day (mg/kg/day) as IV infusion on Days 2-4, and cyclophosphamide at a dose of 250 mg/m^2/day as IV infusion over 15-30 minutes (min) on Days 2-4 in Cycle 1. Then, rituximab at a dose of 500 mg/m^2 as IV infusion on Day 1, cladribine at a dose of 0.12 mg/kg/day as IV infusion on Days 2-4, and cyclophosphamide at a dose of 250 mg/m^2/day as IV infusion over 15-30 min on Days 2-4 were administered in Cycles 2-6. Each cycle was of 28 days in duration.
- Maintenance Arm: Rituximab: Participants received rituximab at a dose of 375 mg/m^2 as IV infusion on Day 1 of Cycle 1 and 500 mg/m^2 as IV infusion on Day 1 of Cycles 2-6, along with cladribine at a dose of 0.12 mg/kg/day as IV infusion on Days 2-4, and cyclophosphamide at a dose of 250 mg/m^2/day as IV infusion over 15-30 min on Days 2-4 of each 28-days cycle for 6 cycles during induction phase. Participants with PR or CR after induction phase who were randomized to maintenance arm received rituximab treatment for 8 cycles. Twelve weeks after the last induction cycle, participants received rituximab at a dose of 375 mg/m^2 as IV infusion on Day 1 of each 12-week cycle until disease progression (up to approximately 96 weeks).
- Observation Arm: No Intervention: Participants received rituximab at a dose of 375 mg/m^2 as IV infusion on Day 1 of Cycle 1 and 500 mg/m^2 as IV infusion on Day 1 of Cycles 2-6, along with cladribine at a dose of 0.12 mg/kg/day as IV infusion on Days 2-4, and cyclophosphamide at a dose of 250 mg/m^2/day as IV infusion over 15-30 min on Days 2-4 of each 28-days cycle for 6 cycles during induction phase. Participants with PR or CR after induction phase who were randomized to observation arm did not receive any intervention. Participants were assessed every 4-weeks for the first 12 weeks and every 12-weeks afterwards up to 96 weeks.
Period: Induction Phase
Arm/Group | Induction: Rituximab, Cladribine, Cyclophosphamide | Maintenance Arm: Rituximab | Observation Arm: No Intervention
Started | 128 | 0 | 0
Completed | 66 | 0 | 0
Not Completed | 62 | 0 | 0
Not completed — Disease Progression | 1 | 0 | 0
Not completed — Eligibility Criteria Violation | 2 | 0 | 0
Not completed — Early Termination - No Additional Info | 59 | 0 | 0
Period: Maintenance/ Observation Phase
Arm/Group | Induction: Rituximab, Cladribine, Cyclophosphamide | Maintenance Arm: Rituximab | Observation Arm: No Intervention
Started | 0 | 33 | 33
Completed | 0 | 5 | 3
Not Completed | 0 | 28 | 30
Not completed — Early Termination - No Additional Info | 0 | 15 | 8
Not completed — Death | 0 | 1 | 2
Not completed — Lost to Follow-up | 0 | 4 | 4
Not completed — Progression | 0 | 5 | 14
Not completed — Relapse | 0 | 3 | 2

BASELINE CHARACTERISTICS:
Population: All enrolled participants who received at least one dose of study medication.
Groups:
- Induction: Rituximab, Cladribine, Cyclophosphamide: Participants received rituximab at a dose of 375 mg/m^2 as IV infusion on Day 1, cladribine at a dose of 0.12 mg/kg/day as IV infusion on Days 2-4, and cyclophosphamide at a dose of 250 mg/m^2/day as IV infusion over 15-30 min on Days 2-4 in Cycle 1. Then, rituximab at a dose of 500 mg/m^2 as IV infusion on Day 1, cladribine at a dose of 0.12 mg/kg/day as IV infusion on Days 2-4, and cyclophosphamide at a dose of 250 mg/m^2/day as IV infusion over 15-30 min on Days 2-4 were administered in Cycles 2-6. Each cycle was of 28 days in duration.
Arm/Group | Induction: Rituximab, Cladribine, Cyclophosphamide
Number analyzed (Participants) | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 84

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Disease Progression (PD), Relapse, or Death Due to Any Cause Assessed According to the National Cancer Institute (NCI) Revised Guidelines for the Diagnosis and Treatment of Chronic Lymphocytic Leukemia (CLL)
Description: PD occurred if any of the following events was observed: appearance of any new lesion, such as enlarged lymph nodes (greater than [>]1.5 centimeters [cm]), splenomegaly, hepatomegaly, or other organ infiltrates; an increase of greater than or equal to (>/=) 50 percent (%) in greatest determined diameter of any previous site; an increase in the previously noted enlargement of the liver or spleen by >/=50%; an increase in the number of blood lymphocytes by >/=50% with B-lymphocytes >/=5000 per microliter (/mcL); transformation to a more aggressive histology; occurrence of cytopenia (neutropenia, anemia, or thrombocytopenia) attributable to CLL.
Time Frame: From randomization to PD, Relapse, or death due to any cause (overall approximately 5 years)
Population: Intent-to-treat (ITT) population included all participants who received at least one dose of study medication and had at least one post-treatment efficacy measurement available. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Groups:
- All Randomized Participants: Participants with PR or CR after induction phase were randomized to observation arm (received no intervention) or to maintenance arm (12 weeks after the last induction cycle, participants received rituximab at a dose of 375 mg/m^2 as IV infusion on Day 1 of each 12-week cycle for 8 cycles or until disease progression [up to approximately 96 weeks]).
Arm/Group | Maintenance Arm: Rituximab | Observation Arm: No Intervention | All Randomized Participants
Number analyzed (Participants) | 33 | 33 | 66
percentage of participants | 27.3 | 54.5 | 40.9

2. Primary Outcome: Progression-Fee Survival (PFS) Assessed According to the NCI Revised Guidelines for the Diagnosis and Treatment of CLL
Description: PFS was defined as the time from date of randomization to date of PD, relapse, or death due to any cause. Participants alive with no evidence of PD or relapse were censored at date of last clinical examination. PD occurred if any of the following events was observed: appearance of any new lesion, such as enlarged lymph nodes (>1.5 cm), splenomegaly, hepatomegaly, or other organ infiltrates; an increase of >/=50% in greatest determined diameter of any previous site; an increase in the previously noted enlargement of the liver or spleen by >/=50%; an increase in the number of blood lymphocytes by >/=50% with B-lymphocytes >/=5000/mcL; transformation to a more aggressive histology; occurrence of cytopenia (neutropenia, anemia, or thrombocytopenia) attributable to CLL.
Time Frame: From randomization to PD, relapse, or death due to any cause (overall approximately 5 years)
Population: ITT population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Maintenance Arm: Rituximab | Observation Arm: No Intervention | All Randomized Participants
Number analyzed (Participants) | 33 | 33 | 66
years | NA [3.0 to NA] — Median and Upper Limit could not be calculated due to insufficient number of participants who had an event. | 2.1 [1.9 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event. | 3.1 [2.2 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
Statistical Analysis 1: Comparison: Maintenance Arm: Rituximab vs Observation Arm: No Intervention; Test type: Superiority; p = 0.028, Log Rank
Statistical Analysis 2: Comparison: Maintenance Arm: Rituximab vs Observation Arm: No Intervention; Univariate comparison; Test type: Superiority; p = 0.033, Cox's proportional hazards regression; Hazard Ratio (HR) = 0.418, 95% CI [0.187 to 0.933]
Statistical Analysis 3: Comparison: Maintenance Arm: Rituximab vs Observation Arm: No Intervention; Multivariate Comparison; Test type: Superiority; p = 0.111, Cox's proportional hazards model; Hazard Ratio (HR) = 0.052, 95% CI 2-sided [0.001 to 1.972]

3. Secondary Outcome: Percentage of Participants With CR or PR Assessed According to the NCI Revised Guidelines for the Diagnosis and Treatment of CLL
Description: CR was achieved if participants met all of the following criteria >/= 2 months after last treatment: no lymphadenopathy (Ly)/ hepatomegaly/ splenomegaly/constitutional symptoms; neutrophils >1500/mcL, platelets (PL) >100,000/mcL, hemoglobin (Hb) >11.0 grams per deciliter (g/dL), bone marrow (BM) sample must be normocellular for age with lymphocytes <30% of nucleated cells. PR: a reduction in Ly (decrease in lymph node size by >/=50% compared to pre-treatment state, no increase in any lymph node, no new enlarged lymph node); a reduction of >/=50% from pre-treatment state in the lymphocytes count, and in enlargement of the spleen or liver; any one of the following: neutrophils >1500/mcL, PL >100,000/mcL (or 50% improvement from baseline), Hb >11.0 g/dL (or 50% improvement from baseline).
Time Frame: 8 weeks after the last dose of rituximab during induction treatment (Week 29) and 12 weeks after the end of maintenance treatment or observation phase (Week 129)
Population: ITT population. Here, 'Overall Number of Participants Analyzed' signifies the number of participants evaluable for this outcome measure and 'Number Analyzed' signifies the number of participants evaluable at specified time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Overall Population: Participants received rituximab at a dose of 375 mg/m^2 as IV infusion on Day 1 of Cycle 1 and 500 mg/m^2 as IV infusion on Day 1 of Cycles 2-6, along with cladribine at a dose of 0.12 mg/kg/day as IV infusion on Days 2-4, and cyclophosphamide at a dose of 250 mg/m^2/day as IV infusion over 15-30 min on Days 2-4 of each 28-days cycle for 6 cycles during induction phase. Participants with PR or CR after induction phase were randomized to observation arm (received no intervention) or to maintenance arm (12 weeks after the last induction cycle, participants received rituximab at a dose of 375 mg/m^2 as IV infusion on Day 1 of each 12-week cycle for 8 cycles or until disease progression [up to approximately 96 weeks]).
Arm/Group | Maintenance Arm: Rituximab | Observation Arm: No Intervention | Overall Population
Number analyzed (Participants) | 21 | 18 | 97
percentage of participants
  Week 29: number analyzed (Participants) | 0 | 0 | 97
  Week 29 |  |  | 73.2 [64.9 to 82.1]
  Week 129: number analyzed (Participants) | 21 | 18 | 39
  Week 129 | 90.5 [85.7 to 100.0] | 72.2 [55.6 to 92.9] | 82.1 [71.8 to 93.5]
Statistical Analysis 1: Comparison: Maintenance Arm: Rituximab vs Observation Arm: No Intervention; Week 129: Univariate Comparison; Test type: Superiority; p = 0.155, Regression, Logistic; Odds Ratio (OR) = 3.654, 95% CI 2-sided [0.674 to 28.337]

4. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) According to Rawstron Criteria in Participants With CR or PR
Description: MRD was defined by the presence of tumor cells in bone marrow, using 4-color flow cytometry of cluster of differentiation (CD)19/CD5/CD20/CD79b. MRD was assessed in participants who achieved CR or PR. CR: if participants met all of the following criteria >/=2 months after last treatment: no Ly/ hepatomegaly/ splenomegaly/constitutional symptoms; neutrophils >1500/mcL, PL >100,000/mcL, Hb >11.0 g/dL, BM sample must be normocellular for age with lymphocytes <30% of nucleated cells. PR: a reduction in Ly; a reduction of >/=50% from pre-treatment state in the lymphocytes count, and in enlargement of the spleen or liver; any one of the following: neutrophils >1500/mcL, PL >100,000/mcL (or 50% improvement from baseline), Hb >11.0 g/dL (or 50% improvement from baseline).
Time Frame: as for outcome 3
Population: as for outcome 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Maintenance Arm: Rituximab | Observation Arm: No Intervention | All Randomized Participants
Number analyzed (Participants) | 14 | 10 | 65
percentage of participants
  Week 29: number analyzed (Participants) | 0 | 0 | 65
  Week 29 |  |  | 15.4 [7.7 to 23.7]
  Week 129: number analyzed (Participants) | 14 | 10 | 24
  Week 129 | 28.6 [14.3 to 55.6] | 20.0 [10.0 to 48.7] | 25.0 [12.5 to 43.9]
Statistical Analysis 1: Comparison: Maintenance Arm: Rituximab vs Observation Arm: No Intervention; Week 129: Univariate comparison; Test type: Superiority; p = 0.634, Regression, Logistic; Odds Ratio (OR) = 0.625, 95% CI 2-sided [0.073 to 4.114]

5. Secondary Outcome: PFS Assessed According to the NCI Revised Guidelines for the Diagnosis and Treatment of CLL According to Clinical and Biochemical Factors
Description: PFS: time from date of randomization to date of PD, relapse, or death from any cause. Participants alive with no evidence of PD or relapse were censored at date of last clinical examination. PD: appearance of any new lesion, such as enlarged lymph nodes (>1.5 cm), splenomegaly, hepatomegaly, or other organ infiltrates; an increase of >/=50% in greatest determined diameter of any previous site; an increase in previously noted enlargement of liver or spleen by >/=50%; an increase in number of blood lymphocytes by >/=50% with B-lymphocytes >/=5000/mcL; transformation to a more aggressive histology; or occurrence of cytopenia attributable to CLL. Rai Stage: staging for CLL, based on lymphocyte, red blood cell and platelet counts and size of lymph nodes, spleen, and liver. Rai Stage I or II are intermediate risk CLL and Rai Stage III or IV are high risk CLL. This outcome measure assessed relationship between clinical markers and clinical outcome (PFS) after study treatment.
Time Frame: From randomization to PD, relapse, or death due to any cause (overall approximately 5 years)
Population: ITT population. Overall Number of Participants Analyzed: participants evaluable for this outcome; Number Analyzed: participants evaluable for specified category. This outcome was planned to be reported for groups defined by clinical and biochemical factors (i.e. reported categories) among All Randomized Participants only.
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 66
years
  Age <60 years: number analyzed (Participants) | 41
  Age <60 years | 3.0 [2.2 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Age >/=60 years: number analyzed (Participants) | 25
  Age >/=60 years | 4.0 [1.9 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Sex: Female: number analyzed (Participants) | 24
  Sex: Female | 4.0 [2.2 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Sex: Male: number analyzed (Participants) | 42
  Sex: Male | 3.0 [2.1 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Rai Stage: I or II: number analyzed (Participants) | 52
  Rai Stage: I or II | 3.1 [2.1 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Rai Stage: III or IV: number analyzed (Participants) | 14
  Rai Stage: III or IV | 3.0 [2.1 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Beta-2-Microglobulin >/= Median Value: number analyzed (Participants) | 27
  Beta-2-Microglobulin >/= Median Value | 1.9 [1.4 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Beta-2-Microglobulin <Median Value: number analyzed (Participants) | 38
  Beta-2-Microglobulin <Median Value | NA [3.5 to NA] — Median and Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Zeta-Associated Protein (ZAP)-70: Negative: number analyzed (Participants) | 45
  Zeta-Associated Protein (ZAP)-70: Negative | 3.0 [2.1 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  ZAP-70 Expression: Positive: number analyzed (Participants) | 15
  ZAP-70 Expression: Positive | NA [4.0 to NA] — Median and Upper Limit could not be calculated due to insufficient number of participants who had an event.
  CD38 Expression: Negative: number analyzed (Participants) | 18
  CD38 Expression: Negative | 2.1 [1.9 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  CD38 Expression: Positive: number analyzed (Participants) | 23
  CD38 Expression: Positive | 2.8 [1.9 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Cytogenetic abnormality 17p: No: number analyzed (Participants) | 54
  Cytogenetic abnormality 17p: No | 3.1 [2.2 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Cytogenetic abnormality 17p: Yes: number analyzed (Participants) | 5
  Cytogenetic abnormality 17p: Yes | 1.9 [1.9 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Cytogenetic abnormality 13q: No: number analyzed (Participants) | 21
  Cytogenetic abnormality 13q: No | 3.5 [1.4 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Cytogenetic abnormality 13q: Yes: number analyzed (Participants) | 31
  Cytogenetic abnormality 13q: Yes | 3.0 [1.9 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Cytogenetic abnormality 11q: No: number analyzed (Participants) | 37
  Cytogenetic abnormality 11q: No | 3.5 [2.1 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Cytogenetic abnormality 11q: Yes: number analyzed (Participants) | 18
  Cytogenetic abnormality 11q: Yes | 2.8 [1.9 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Cytogenetic abnormality 12q: No: number analyzed (Participants) | 41
  Cytogenetic abnormality 12q: No | 2.2 [1.9 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
  Cytogenetic abnormality 12q: Yes: number analyzed (Participants) | 4
  Cytogenetic abnormality 12q: Yes | 3.1 [3.1 to NA] — Upper Limit could not be calculated due to insufficient number of participants who had an event.
Statistical Analysis 1: Comparison: All Randomized Participants; Multivariate Comparison: Age <60 years versus Age >/=60 years; Test type: Superiority; p = 0.752, Cox's proportional hazards model; Hazard Ratio (HR) = 0.769, 95% CI 2-sided [0.151 to 3.920]
Statistical Analysis 2: Comparison: All Randomized Participants; Multivariate Comparison: Sex: Female versus Male; Test type: Superiority; p = 0.128, Cox's proportional hazards model; Hazard Ratio (HR) = 0.068, 95% CI 2-sided [0.002 to 2.158]
Statistical Analysis 3: Comparison: All Randomized Participants; Multivariate Comparison: Rai Stage: I or II versus Rai Stage: III or IV; Test type: Superiority; p = 0.728, Cox's proportional hazards model; Hazard Ratio (HR) = 2.282, 95% CI 2-sided [0.022 to 240.864]
Statistical Analysis 4: Comparison: All Randomized Participants; Multivariate Comparison: Beta-2-Microglobulin >/= Median Value versus Beta-2-Microglobulin <Median Value; Test type: Superiority; p = 0.048, Cox's proportional hazards model; Hazard Ratio (HR) = 26.275, 95% CI 2-sided [1.036 to 666.708]
Statistical Analysis 5: Comparison: All Randomized Participants; Multivariate Comparison: ZAP-70 Expression Negative versus Positive; Test type: Superiority; p = 0.417, Cox's proportional hazards model; Hazard Ratio (HR) = 0.210, 95% CI 2-sided [0.005 to 9.100]
Statistical Analysis 6: Comparison: All Randomized Participants; Multivariate Comparison: CD38 Expression Negative versus Positive; Test type: Superiority; p = 0.134, Cox's proportional hazards model; Hazard Ratio (HR) = 0.197, 95% CI 2-sided [0.024 to 1.647]
Statistical Analysis 7: Comparison: All Randomized Participants; Multivariate Comparison: Cytogenetic abnormality 17p No versus Yes; Test type: Superiority; p = 0.426, Cox's proportional hazards model; Hazard Ratio (HR) = 8.373, 95% CI 2-sided [0.045 to 1568.717]
Statistical Analysis 8: Comparison: All Randomized Participants; Multivariate Comparison: Cytogenetic abnormality 13q No versus Yes; Test type: Superiority; p = 0.733, Cox's proportional hazards model; Hazard Ratio (HR) = 0.438, 95% CI 2-sided [0.004 to 50.334]
Statistical Analysis 9: Comparison: All Randomized Participants; Multivariate Comparison: Cytogenetic abnormality 11q No versus Yes; Test type: Superiority; p = 0.463, Cox's proportional hazards model; Hazard Ratio (HR) = 2.621, 95% CI 2-sided [0.200 to 34.422]
Statistical Analysis 10: Comparison: All Randomized Participants; Multivariate Comparison: Cytogenetic abnormality 12q No versus Yes; Test type: Superiority; p = 0.397, Cox's proportional hazards model; Hazard Ratio (HR) = 0.288, 95% CI 2-sided [0.016 to 5.122]

6. Secondary Outcome: Percentage of Participants With CR or PR Assessed According to the NCI Revised Guidelines for the Diagnosis and Treatment of CLL According to Clinical and Biochemical Factors at Week 29
Description: CR was achieved if participants met all of the following criteria >/= 2 months after last treatment: no Ly/ hepatomegaly/ splenomegaly/constitutional symptoms; neutrophils >1500/mcL, PL >100,000/mcL, Hb >11.0 g/dL, BM sample must be normocellular for age with lymphocytes <30% of nucleated cells. PR: a reduction in Ly; a reduction of >/=50% from pre-treatment state in the lymphocytes count, and in enlargement of the spleen or liver; any one of the following: neutrophils >1500/mcL, PL >100,000/mcL (or 50% improvement from baseline), Hb >11.0 g/dL (or 50% improvement from baseline). Rai Stage: staging for CLL, based on lymphocyte, red blood cell and platelet counts and size of lymph nodes, spleen, and liver. Rai Stage I or II are intermediate risk CLL and Rai Stage III or IV are high risk CLL. This outcome measure assessed the relationship between clinical markers and clinical outcome (response) after study treatment.
Time Frame: 8 weeks after the last dose of rituximab during induction treatment (Week 29)
Population: ITT population. Number Analyzed: participants evaluable for specified category. This outcome was planned to be reported for groups defined by clinical and biochemical factors (i.e. reported categories) among Participants included in Overall IIT population only.
Measure: Number; unit: percentage of participants
Arm/Group | Overall Population
Number analyzed (Participants) | 97
percentage of participants
  Age <60 years: number analyzed (Participants) | 60
  Age <60 years | 73.3
  Age >/=60 years: number analyzed (Participants) | 37
  Age >/=60 years | 73.0
  Sex: Female: number analyzed (Participants) | 31
  Sex: Female | 80.6
  Sex: Male: number analyzed (Participants) | 66
  Sex: Male | 69.7
  Rai Stage: I or II: number analyzed (Participants) | 71
  Rai Stage: I or II | 77.5
  Rai Stage: III or IV: number analyzed (Participants) | 26
  Rai Stage: III or IV | 61.5
  Beta-2-Microglobulin >/= Median Value: number analyzed (Participants) | 48
  Beta-2-Microglobulin >/= Median Value | 64.6
  Beta-2-Microglobulin <Median Value: number analyzed (Participants) | 47
  Beta-2-Microglobulin <Median Value | 83.0
  ZAP-70 Expression: Negative: number analyzed (Participants) | 70
  ZAP-70 Expression: Negative | 67.1
  ZAP-70 Expression: Positive: number analyzed (Participants) | 19
  ZAP-70 Expression: Positive | 94.7
  CD38 Expression: Negative: number analyzed (Participants) | 26
  CD38 Expression: Negative | 73.1
  CD38 Expression: Positive: number analyzed (Participants) | 35
  CD38 Expression: Positive | 71.4
  Cytogenetic abnormality 17p: No: number analyzed (Participants) | 81
  Cytogenetic abnormality 17p: No | 72.8
  Cytogenetic abnormality 17p: Yes: number analyzed (Participants) | 7
  Cytogenetic abnormality 17p: Yes | 71.4
  Cytogenetic abnormality 13q: No: number analyzed (Participants) | 35
  Cytogenetic abnormality 13q: No | 62.9
  Cytogenetic abnormality 13q: Yes: number analyzed (Participants) | 46
  Cytogenetic abnormality 13q: Yes | 76.1
  Cytogenetic abnormality 11q: No: number analyzed (Participants) | 59
  Cytogenetic abnormality 11q: No | 69.5
  Cytogenetic abnormality 11q: Yes: number analyzed (Participants) | 24
  Cytogenetic abnormality 11q: Yes | 79.2
  Cytogenetic abnormality 12q: No: number analyzed (Participants) | 68
  Cytogenetic abnormality 12q: No | 67.6
  Cytogenetic abnormality 12q: Yes: number analyzed (Participants) | 6
  Cytogenetic abnormality 12q: Yes | 66.7
Statistical Analysis 1: Comparison: Overall Population; Univariate Comparison: Age <60 years versus Age >/=60 years; Test type: Superiority; p = 0.969, Regression, Logistic; Odds Ratio (OR) = 0.982, 95% CI 2-sided [0.393 to 2.531]
Statistical Analysis 2: Comparison: Overall Population; Univariate Comparison: Sex: Female versus Male; Test type: Superiority; p = 0.260, Regression, Logistic; Odds Ratio (OR) = 0.552, 95% CI 2-sided [0.183 to 1.488]
Statistical Analysis 3: Comparison: Overall Population; Univariate Comparison: Rai Stage: I or II versus Rai Stage: III or IV; Test type: Superiority; p = 0.121, Regression, Logistic; Odds Ratio (OR) = 0.465, 95% CI 2-sided [0.177 to 1.242]
Statistical Analysis 4: Comparison: Overall Population; Univariate Comparison: Beta-2-Microglobulin >/= Median Value versus Beta-2-Microglobulin <Median Value; Test type: Superiority; p = 0.045, Regression, Logistic; Odds Ratio (OR) = 0.374, 95% CI 2-sided [0.137 to 0.957]
Statistical Analysis 5: Comparison: Overall Population; Univariate Comparison: ZAP-70 Expression Negative versus Positive; Test type: Superiority; p = 0.040, Regression, Logistic; Odds Ratio (OR) = 8.809, 95% CI 2-sided [1.655 to 163.316]
Statistical Analysis 6: Comparison: Overall Population; Univariate Comparison: CD38 Expression Negative versus Positive; Test type: Superiority; p = 0.887, Regression, Logistic; Odds Ratio (OR) = 0.921, 95% CI 2-sided [0.287 to 2.851]
Statistical Analysis 7: Comparison: Overall Population; Univariate Comparison: Cytogenetic abnormality 17p No versus Yes; Test type: Superiority; p = 0.936, Regression, Logistic; Odds Ratio (OR) = 0.932, 95% CI 2-sided [0.186 to 6.839]
Statistical Analysis 8: Comparison: Overall Population; Univariate Comparison: Cytogenetic abnormality 13q No versus Yes; Test type: Superiority; p = 0.199, Regression, Logistic; Odds Ratio (OR) = 1.880, 95% CI 2-sided [0.719 to 5.012]
Statistical Analysis 9: Comparison: Overall Population; Univariate Comparison: Cytogenetic abnormality 11q No versus Yes; Test type: Superiority; p = 0.375, Regression, Logistic; Odds Ratio (OR) = 1.668, 95% CI 2-sided [0.566 to 5.649]
Statistical Analysis 10: Comparison: Overall Population; Univariate Comparison: Cytogenetic abnormality 12q No versus Yes; Test type: Superiority; p = 0.961, Regression, Logistic; Odds Ratio (OR) = 0.957, 95% CI 2-sided [0.173 to 7.275]

7. Secondary Outcome: Percentage of Participants With CR or PR Assessed According to the NCI Revised Guidelines for the Diagnosis and Treatment of CLL According to Clinical and Biochemical Factors at Week 129
Description: CR was achieved if participants met all of the following criteria >/=2 months after last treatment: no Ly/ hepatomegaly/ splenomegaly/constitutional symptoms; neutrophils >1500/mcL, PL >100,000/mcL, Hb >11.0 g/dL, BM sample must be normocellular for age with lymphocytes <30% of nucleated cells. PR: a reduction in Ly; a reduction of >/=50% from pre-treatment state in the lymphocytes count, and in enlargement of the spleen or liver; any one of the following: neutrophils >1500/mcL, PL >100,000/mcL (or 50% improvement from baseline), Hb >11.0 g/dL (or 50% improvement from baseline). Rai Stage: staging for CLL, based on lymphocyte, red blood cell and platelet counts and size of lymph nodes, spleen, and liver. Rai Stage I or II are intermediate risk CLL and Rai Stage III or IV are high risk CLL. This outcome measure assessed the relationship between clinical markers and clinical outcome (response) after study treatment.
Time Frame: 12 weeks after the end of maintenance treatment or observation phase (Week 129)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 39
percentage of participants
  Age <60 years: number analyzed (Participants) | 26
  Age <60 years | 80.8
  Age >/=60 years: number analyzed (Participants) | 13
  Age >/=60 years | 84.6
  Sex: Female: number analyzed (Participants) | 14
  Sex: Female | 85.7
  Sex: Male: number analyzed (Participants) | 25
  Sex: Male | 80.0
  Rai Stage: I or II: number analyzed (Participants) | 31
  Rai Stage: I or II | 80.6
  Rai Stage: III or IV: number analyzed (Participants) | 8
  Rai Stage: III or IV | 87.5
  Beta-2-Microglobulin >/= Median Value: number analyzed (Participants) | 13
  Beta-2-Microglobulin >/= Median Value | 76.9
  Beta-2-Microglobulin <Median Value: number analyzed (Participants) | 25
  Beta-2-Microglobulin <Median Value | 84.0
  ZAP-70 Expression: Negative: number analyzed (Participants) | 24
  ZAP-70 Expression: Negative | 83.3
  ZAP-70 Expression: Positive: number analyzed (Participants) | 12
  ZAP-70 Expression: Positive | 83.3
  CD38 Expression: Negative: number analyzed (Participants) | 9
  CD38 Expression: Negative | 77.8
  CD38 Expression: Positive: number analyzed (Participants) | 12
  CD38 Expression: Positive | 75.0
  Cytogenetic abnormality 17p: No: number analyzed (Participants) | 30
  Cytogenetic abnormality 17p: No | 86.7
  Cytogenetic abnormality 17p: Yes: number analyzed (Participants) | 2
  Cytogenetic abnormality 17p: Yes | 50.0
  Cytogenetic abnormality 13q: No: number analyzed (Participants) | 10
  Cytogenetic abnormality 13q: No | 90.0
  Cytogenetic abnormality 13q: Yes: number analyzed (Participants) | 17
  Cytogenetic abnormality 13q: Yes | 76.5
  Cytogenetic abnormality 11q: No: number analyzed (Participants) | 19
  Cytogenetic abnormality 11q: No | 84.2
  Cytogenetic abnormality 11q: Yes: number analyzed (Participants) | 10
  Cytogenetic abnormality 11q: Yes | 80.0
  Cytogenetic abnormality 12q: No: number analyzed (Participants) | 21
  Cytogenetic abnormality 12q: No | 76.2
  Cytogenetic abnormality 12q: Yes: number analyzed (Participants) | 3
  Cytogenetic abnormality 12q: Yes | 100.0
Statistical Analysis 1: Comparison: All Randomized Participants; Univariate Comparison: Age <60 years versus Age >/=60 years; Test type: Superiority; p = 0.768, Regression, Logistic; Odds Ratio (OR) = 1.310, 95% CI 2-sided [0.237 to 10.189]
Statistical Analysis 2: Comparison: All Randomized Participants; Univariate Comparison: Sex: Female versus Male; Test type: Superiority; p = 0.657, Regression, Logistic; Odds Ratio (OR) = 0.667, 95% CI 2-sided [0.086 to 3.653]
Statistical Analysis 3: Comparison: All Randomized Participants; Univariate Comparison: Rai Stage: I or II versus Rai Stage: III or IV; Test type: Superiority; p = 0.655, Regression, Logistic; Odds Ratio (OR) = 1.680, 95% CI 2-sided [0.229 to 34.486]
Statistical Analysis 4: Comparison: All Randomized Participants; Univariate Comparison: Beta-2-Microglobulin >/= Median Value versus Beta-2-Microglobulin <Median Value; Test type: Superiority; p = 0.595, Regression, Logistic; Odds Ratio (OR) = 0.635, 95% CI 2-sided [0.117 to 3.730]
Statistical Analysis 5: Comparison: All Randomized Participants; Univariate Comparison: ZAP-70 Expression Negative versus Positive; Test type: Superiority; p = 1.000, Regression, Logistic; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.164 to 8.102]
Statistical Analysis 6: Comparison: All Randomized Participants; Univariate Comparison: CD38 Expression Negative versus Positive; Test type: Superiority; p = 0.882, Regression, Logistic; Odds Ratio (OR) = 0.857, 95% CI 2-sided [0.093 to 6.636]
Statistical Analysis 7: Comparison: All Randomized Participants; Univariate Comparison: Cytogenetic abnormality 17p No versus Yes; Test type: Superiority; p = 0.216, Regression, Logistic; Odds Ratio (OR) = 0.154, 95% CI 2-sided [0.005 to 4.405]
Statistical Analysis 8: Comparison: All Randomized Participants; Univariate Comparison: Cytogenetic abnormality 13q No versus Yes; Test type: Superiority; p = 0.396, Regression, Logistic; Odds Ratio (OR) = 0.361, 95% CI 2-sided [0.017 to 2.971]
Statistical Analysis 9: Comparison: All Randomized Participants; Univariate Comparison: Cytogenetic abnormality 11q No versus Yes; Test type: Superiority; p = 0.776, Regression, Logistic; Odds Ratio (OR) = 0.750, 95% CI 2-sided [0.103 to 6.572]

8. Secondary Outcome: Percentage of Participants With MRD According to Rawstron Criteria in Participants With CR or PR According to Clinical and Biochemical Factors at Week 29
Description: MRD: the presence of tumor cells in bone marrow, using 4-color flow cytometry of CD19/CD5/CD20/CD79b. MRD was assessed in participants who achieved CR or PR. CR (>/=2 months after last treatment): no Ly/ hepatomegaly/ splenomegaly/constitutional symptoms; neutrophils >1500/mcL, PL >100,000/mcL, Hb >11.0 g/dL, BM sample must be normocellular for age with lymphocytes <30% of nucleated cells. PR: a reduction in Ly; a reduction of >/=50% from pre-treatment state in the lymphocytes count, and in enlargement of the spleen or liver; any one of the following: neutrophils >1500/mcL, PL >100,000/mcL (or 50% improvement from baseline), Hb >11.0 g/dL (or 50% improvement from baseline). Rai Stage: staging for CLL, based on lymphocyte, red blood cell and platelet counts and size of lymph nodes, spleen, and liver. Rai Stage I or II are intermediate risk CLL and Rai Stage III or IV are high risk CLL. This outcome measure assessed relationship between clinical markers and MRD after study treatment.
Time Frame: 8 weeks after the last dose of rituximab during induction treatment (Week 29)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Groups:
- All Randomized Participants: Participants with PR or CR after induction phase were randomized to either observation arm (received no intervention) or to maintenance arm (received maintenance treatment with rituximab administered at a dose of 375 mg/m^2 as IV infusion on Day 1 of each 12-week cycle for 8 cycles until disease progression for up to approximately 96 weeks).
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 65
percentage of participants
  Age <60 years: number analyzed (Participants) | 41
  Age <60 years | 87.8
  Age >/=60 years: number analyzed (Participants) | 24
  Age >/=60 years | 79.2
  Sex: Female: number analyzed (Participants) | 24
  Sex: Female | 87.5
  Sex: Male: number analyzed (Participants) | 41
  Sex: Male | 82.9
  Rai Stage: I or II: number analyzed (Participants) | 51
  Rai Stage: I or II | 80.4
  Rai Stage: III or IV: number analyzed (Participants) | 14
  Rai Stage: III or IV | 100.0
  Beta-2-Microglobulin >/= Median Value: number analyzed (Participants) | 29
  Beta-2-Microglobulin >/= Median Value | 93.1
  Beta-2-Microglobulin <Median Value: number analyzed (Participants) | 35
  Beta-2-Microglobulin <Median Value | 77.1
  ZAP-70 Expression: Negative: number analyzed (Participants) | 46
  ZAP-70 Expression: Negative | 82.6
  ZAP-70 Expression: Positive: number analyzed (Participants) | 15
  ZAP-70 Expression: Positive | 100.0
  CD38 Expression: Negative: number analyzed (Participants) | 18
  CD38 Expression: Negative | 83.3
  CD38 Expression: Positive: number analyzed (Participants) | 22
  CD38 Expression: Positive | 95.5
  Cytogenetic abnormality 17p: No: number analyzed (Participants) | 55
  Cytogenetic abnormality 17p: No | 83.6
  Cytogenetic abnormality 17p: Yes: number analyzed (Participants) | 4
  Cytogenetic abnormality 17p: Yes | 100.0
  Cytogenetic abnormality 13q: No: number analyzed (Participants) | 19
  Cytogenetic abnormality 13q: No | 84.2
  Cytogenetic abnormality 13q: Yes: number analyzed (Participants) | 33
  Cytogenetic abnormality 13q: Yes | 81.8
  Cytogenetic abnormality 11q: No: number analyzed (Participants) | 36
  Cytogenetic abnormality 11q: No | 83.3
  Cytogenetic abnormality 11q: Yes: number analyzed (Participants) | 19
  Cytogenetic abnormality 11q: Yes | 84.2
  Cytogenetic abnormality 12q: No: number analyzed (Participants) | 41
  Cytogenetic abnormality 12q: No | 80.5
  Cytogenetic abnormality 12q: Yes: number analyzed (Participants) | 4
  Cytogenetic abnormality 12q: Yes | 75.0
Statistical Analysis 1: Comparison: All Randomized Participants; Univariate Comparison: Age <60 years versus Age >/=60 years; Test type: Superiority; p = 0.357, Regression, Logistic; Odds Ratio (OR) = 0.528, 95% CI 2-sided [0.131 to 2.114]
Statistical Analysis 2: Comparison: All Randomized Participants; Univariate Comparison: Sex: Female versus Male; Test type: Superiority; p = 0.623, Regression, Logistic; Odds Ratio (OR) = 0.694, 95% CI 2-sided [0.138 to 2.800]
Statistical Analysis 3: Comparison: All Randomized Participants; Univariate Comparison: Beta-2-Microglobulin >/= Median Value versus Beta-2-Microglobulin <Median Value; Test type: Superiority; p = 0.097, Regression, Logistic; Odds Ratio (OR) = 4.000, 95% CI 2-sided [0.901 to 28.158]
Statistical Analysis 4: Comparison: All Randomized Participants; Univariate Comparison: CD38 Expression Negative versus Positive; Test type: Superiority; p = 0.233, Regression, Logistic; Odds Ratio (OR) = 4.200, 95% CI 2-sided [0.484 to 89.588]
Statistical Analysis 5: Comparison: All Randomized Participants; Univariate Comparison: Cytogenetic abnormality 13q No versus Yes; Test type: Superiority; p = 0.826, Regression, Logistic; Odds Ratio (OR) = 0.844, 95% CI 2-sided [0.161 to 3.681]
Statistical Analysis 6: Comparison: All Randomized Participants; Univariate Comparison: Cytogenetic abnormality 11q No versus Yes; Test type: Superiority; p = 0.933, Regression, Logistic; Odds Ratio (OR) = 1.067, 95% CI 2-sided [0.246 to 5.581]
Statistical Analysis 7: Comparison: All Randomized Participants; Univariate Comparison: Cytogenetic abnormality 12q No versus Yes; Test type: Superiority; p = 0.794, Regression, Logistic; Odds Ratio (OR) = 0.727, 95% CI 2-sided [0.080 to 15.779]

9. Secondary Outcome: Percentage of Participants With MRD According to Rawstron Criteria in Participants With CR or PR According to Clinical and Biochemical Factors at Week 129
Description: as for outcome 8
Time Frame: 12 weeks after the end of maintenance treatment or observation phase (Week 129)
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | All Randomized Participants
Number analyzed (Participants) | 24
percentage of participants
  Age <60 years: number analyzed (Participants) | 18
  Age <60 years | 72.2
  Age >/=60 years: number analyzed (Participants) | 6
  Age >/=60 years | 83.3
  Sex: Female: number analyzed (Participants) | 7
  Sex: Female | 71.4
  Sex: Male: number analyzed (Participants) | 17
  Sex: Male | 76.5
  Rai Stage: I or II: number analyzed (Participants) | 20
  Rai Stage: I or II | 75.0
  Rai Stage: III or IV: number analyzed (Participants) | 4
  Rai Stage: III or IV | 75.0
  Beta-2-Microglobulin >/= Median Value: number analyzed (Participants) | 9
  Beta-2-Microglobulin >/= Median Value | 88.9
  Beta-2-Microglobulin <Median Value: number analyzed (Participants) | 14
  Beta-2-Microglobulin <Median Value | 71.4
  ZAP-70 Expression: Negative: number analyzed (Participants) | 15
  ZAP-70 Expression: Negative | 66.7
  ZAP-70 Expression: Positive: number analyzed (Participants) | 7
  ZAP-70 Expression: Positive | 100.0
  CD38 Expression: Negative: number analyzed (Participants) | 5
  CD38 Expression: Negative | 60.0
  CD38 Expression: Positive: number analyzed (Participants) | 9
  CD38 Expression: Positive | 77.8
  Cytogenetic abnormality 17p: No: number analyzed (Participants) | 21
  Cytogenetic abnormality 17p: No | 76.2
  Cytogenetic abnormality 17p: Yes: number analyzed (Participants) | 1
  Cytogenetic abnormality 17p: Yes | 0.0
  Cytogenetic abnormality 13q: No: number analyzed (Participants) | 8
  Cytogenetic abnormality 13q: No | 75.0
  Cytogenetic abnormality 13q: Yes: number analyzed (Participants) | 12
  Cytogenetic abnormality 13q: Yes | 66.7
  Cytogenetic abnormality 11q: No: number analyzed (Participants) | 12
  Cytogenetic abnormality 11q: No | 66.7
  Cytogenetic abnormality 11q: Yes: number analyzed (Participants) | 8
  Cytogenetic abnormality 11q: Yes | 75.0
  Cytogenetic abnormality 12q: No: number analyzed (Participants) | 15
  Cytogenetic abnormality 12q: No | 66.7
  Cytogenetic abnormality 12q: Yes: number analyzed (Participants) | 3
  Cytogenetic abnormality 12q: Yes | 66.7
Statistical Analysis 1: Comparison: All Randomized Participants; Univariate Comparison: Age <60 years versus Age >/=60 years; Test type: Superiority; p = 0.591, Regression, Logistic; Odds Ratio (OR) = 1.923, 95% CI 2-sided [0.225 to 41.751]
Statistical Analysis 2: Comparison: All Randomized Participants; Univariate Comparison: Sex: Female versus Male; Test type: Superiority; p = 0.796, Regression, Logistic; Odds Ratio (OR) = 1.300, 95% CI 2-sided [0.147 to 9.222]
Statistical Analysis 3: Comparison: All Randomized Participants; Univariate Comparison: Beta-2-Microglobulin >/= Median Value versus Beta-2-Microglobulin <Median Value; Test type: Superiority; p = 0.338, Regression, Logistic; Odds Ratio (OR) = 3.200, 95% CI 2-sided [0.375 to 69.479]
Statistical Analysis 4: Comparison: All Randomized Participants; Univariate Comparison: CD38 Expression Negative versus Positive; Test type: Superiority; p = 0.486, Regression, Logistic; Odds Ratio (OR) = 2.333, 95% CI 2-sided [0.201 to 29.008]
Statistical Analysis 5: Comparison: All Randomized Participants; Univariate Comparison: Cytogenetic abnormality 13q No versus Yes; Test type: Superiority; p = 0.691, Regression, Logistic; Odds Ratio (OR) = 0.667, 95% CI 2-sided [0.074 to 4.722]
Statistical Analysis 6: Comparison: All Randomized Participants; Univariate Comparison: Cytogenetic abnormality 11q No versus Yes; Test type: Superiority; p = 0.691, Regression, Logistic; Odds Ratio (OR) = 1.500, 95% CI 2-sided [0.212 to 13.563]
Statistical Analysis 7: Comparison: All Randomized Participants; Univariate Comparison: Cytogenetic abnormality 12q No versus Yes; Test type: Superiority; p = 1.000, Regression, Logistic; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.076 to 24.621]
Statistical Analysis 8: Comparison: All Randomized Participants; Univariate Comparison: Rai Stage: I or II versus Rai Stage: III or IV; Test type: Superiority; p = 1.000, Regression, Logistic; Odds Ratio (OR) = 1.000, 95% CI 2-sided [0.099 to 22.791]

ADVERSE EVENTS:
Time Frame: From Day 1 to end of study (up to 261 weeks)
Description: All enrolled participants who received at least one dose of study medication were included in the analysis.
Groups:
- Induction (Excluding Maintenance/ Observation): Participants received rituximab at a dose of 375 mg/m^2 as IV infusion on Day 1, cladribine at a dose of 0.12 mg/kg/day as IV infusion on Days 2-4, and cyclophosphamide at a dose of 250 mg/m^2/day as IV infusion over 15-30 min on Days 2-4 in Cycle 1. Then, rituximab at a dose of 500 mg/m^2 as IV infusion on Day 1, cladribine at a dose of 0.12 mg/kg/day as IV infusion on Days 2-4, and cyclophosphamide at a dose of 250 mg/m^2/day as IV infusion over 15-30 min on Days 2-4 were administered in Cycles 2-6. Each cycle was of 28 days in duration. Only participants who were not randomized to maintenance or observation arm were included.
- All Participants: All enrolled participants who received at least one dose of study medication were included in the analysis.
Arm/Group | Induction (Excluding Maintenance/ Observation) | Maintenance Arm: Rituximab | Observation Arm: No Intervention | All Participants
Serious Adverse Events (participants affected / at risk) | 23/62 | 13/33 | 9/33 | 45/128
Other Adverse Events (participants affected / at risk) | 58/62 | 31/33 | 32/33 | 121/128
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Induction (Excluding Maintenance/ Observation) (N=62) | Maintenance Arm: Rituximab (N=33) | Observation Arm: No Intervention (N=33) | All Participants (N=128)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 2
Aplasia pure red cell (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 2 | 0 | 6
Leukopenia (Blood and lymphatic system disorders) | 0 | 1 | 2 | 3
Neutropenia (Blood and lymphatic system disorders) | 1 | 4 | 0 | 5
Pancytopenia (Blood and lymphatic system disorders) | 3 | 0 | 0 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Disease progression (General disorders) | 0 | 0 | 1 | 1
Pelvic mass (General disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 1
Soft tissue inflammation (General disorders) | 0 | 1 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Appendiceal abscess (Infections and infestations) | 1 | 0 | 0 | 1
Bacterial sepsis (Infections and infestations) | 1 | 0 | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 2 | 0 | 0 | 2
Herpes zoster (Infections and infestations) | 2 | 0 | 1 | 3
Oral fungal infection (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 1 | 1 | 2 | 4
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Abnormal loss of weight (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Groin abscess (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Myositis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Sympathetic posterior cervical syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Acute leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Breast cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Lip neoplasm malignant stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Richter's syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 2
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 1 | 1
Loss of consciousness (Nervous system disorders) | 1 | 0 | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 0 | 1 | 1
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Uterine polyp (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Acne varioliformis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Cellulitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Toxic epidermal necrolysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Heart valve operation (Surgical and medical procedures) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Induction (Excluding Maintenance/ Observation) (N=62) | Maintenance Arm: Rituximab (N=33) | Observation Arm: No Intervention (N=33) | All Participants (N=128)
Anaemia (Blood and lymphatic system disorders) | 11 | 1 | 3 | 15
Leukopenia (Blood and lymphatic system disorders) | 1 | 6 | 6 | 13
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3 | 5 | 8
Neutropenia (Blood and lymphatic system disorders) | 47 | 26 | 20 | 93
Thrombocytopenia (Blood and lymphatic system disorders) | 18 | 5 | 5 | 28
Cardiomegaly (Cardiac disorders) | 0 | 2 | 0 | 2
Goitre (Endocrine disorders) | 0 | 1 | 2 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 2 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 2 | 3
Diarrhoea (Gastrointestinal disorders) | 6 | 7 | 3 | 16
Nausea (Gastrointestinal disorders) | 7 | 12 | 4 | 23
Vomiting (Gastrointestinal disorders) | 4 | 0 | 1 | 5
Asthenia (General disorders) | 3 | 2 | 2 | 7
Chills (General disorders) | 8 | 3 | 3 | 14
Influenza like illness (General disorders) | 0 | 0 | 2 | 2
Pyrexia (General disorders) | 11 | 5 | 3 | 19
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 3 | 3
Hepatic steatosis (Hepatobiliary disorders) | 0 | 2 | 2 | 4
Chronic sinusitis (Infections and infestations) | 0 | 2 | 0 | 2
Oral herpes (Infections and infestations) | 2 | 1 | 2 | 5
Respiratory tract infection (Infections and infestations) | 1 | 2 | 2 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 3 | 6 | 13
Urinary tract infection (Infections and infestations) | 0 | 3 | 1 | 4
Blood lactate dehydrogenase increased (Investigations) | 1 | 0 | 2 | 3
Hepatic enzyme increased (Investigations) | 0 | 2 | 2 | 4
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 0 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 5 | 4 | 2 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 | 4
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 2
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2 | 1 | 3
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 3 | 3 | 6
Headache (Nervous system disorders) | 2 | 2 | 2 | 6
Sciatica (Nervous system disorders) | 1 | 2 | 1 | 4
Nephroptosis (Renal and urinary disorders) | 0 | 0 | 3 | 3
Renal cyst (Renal and urinary disorders) | 0 | 2 | 5 | 7
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 2 | 0 | 2
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 3 | 1 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 0 | 6
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 4 | 7
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 4
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 6 | 2 | 8
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 3 | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 1 | 4
Rash pruritic (Skin and subcutaneous tissue disorders) | 4 | 1 | 1 | 6
Aortic arteriosclerosis (Vascular disorders) | 0 | 1 | 2 | 3
Hypertension (Vascular disorders) | 2 | 4 | 3 | 9
Hypotension (Vascular disorders) | 3 | 0 | 2 | 5

LIMITATIONS AND CAVEATS:
In 2011 the recruitment was stopped due to low enrollment rate, and in 2015 the trial was prematurely discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.